CLINICAL TRIAL: NCT03589222
Title: An Open-label, Multicenter, Phase 2 Trial of Selinexor (KPT-330), Bortezomib and Low-dose Dexamethasone Plus Daratumumab (SELIBORDARA) for the Treatment of Patients With Refractory or Relapsed and Refractory Multiple Myeloma
Brief Title: SELIBORDARA: Selinexor, Bortezomib and Daratumumab in Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM- SELIBORDARA
Record Dates: First submitted 2018-06-12; First posted 2018-07-17 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor; daratumumab; Bortezomib; Dexamethasone

STUDY DESIGN:
Intervention Model Description: This is an investigator-sponsored, open-label, non-randomized Phase 2 study to evaluate the efficacy and safety of this combination for a total of 62 patients with refractory or relapsed/refractory MM patients. The treatment will be given until progression of the disease or inacceptable toxicity. This trial will be conducted in approximately 15-centers in Spain
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selinexor, Daratumumab, Bortezomib and dexamethasone (Experimental): Selinexor will be administered via oral at flat dose of 100 mg weekly in 4 out of each 4-week cycle plus dexamethasone 40 or 20 mg mg orally with each dose of selinexor in combination with daratumumab at dose of 16 mg/Kg iv weekly on days 1, 8, 15 and 22 during the first two cycles; on days 1 and 15 (Q2W) during the cycles 3 to 6; and on day 1 (Q4W) thereafter and bortezomib will be given via subcutaneous at dose of 1.3 mg/m2 on days 1, 8, 15 and 22 starting from the first cycle and on days 1 and 15 (Q2W) since cycle 9. Each cycle is of 4 weeks of duration
  Interventions: Drug: Selinexor; Drug: Daratumumab; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — Selinexor will be administered via oral at flat dose of 100 mg weekly in 4 out of each 4-week cycle
Drug: Daratumumab — daratumumab at dose of 16 mg/Kg iv weekly on days 1, 8, 15 and 22 during the first two cycles; on days 1 and 15 (Q2W) during the cycles 3 to 6; and on day 1 (Q4W) thereafter
Drug: Bortezomib — bortezomib will be given via subcutaneous at dose of 1.3 mg/m2 on days 1, 8, 15 and 22 starting from the first cycle and on days 1 and 15 (Q2W) since cycle 9
Drug: Dexamethasone — dexamethasone is 20mg (IV) when given on days that daratumumab is administered (as pre-infusion medication) plus 20 mg of dexamethasone (VO) the day after and the dose of dexamethasone is 40mg (VO) on days when daratumumab is not administered

SUMMARY:
Phase 2, single-arm, open, non-randomized, multicenter study of the SINE™ compound selinexor plus low-dose dexamethasone, in combination with bortezomib and daratumumab.

100 mg selinexor (on days 1, 8, 15 and 22), plus 40 mg dexamethasone (20 mg IV the day of daratumumab and selinexor and 20 mg oral administration the day after daratumumab and selinexor) both weekly as continuous therapy.

Bortezomib will be given via subcutaneous at dose of 1.3 mg/m2 once weekly on days 1, 8, 15 and 22 during the cycles 1 to cycle 8, and on day 1 and day 15 of each cycle thereafter as continuous therapy.

Daratumumab will be given via intravenous at dose of 16 mg/Kg on days 1, 8, 15 and 22 (weekly) during the cycles 1 and 2, every two weeks (on days 1 and 15) during the cycles 3 to 6 and on day 1 of each cycle thereafter as continuous therapy.

Patients may continue indefinitely and there is no maximum treatment duration

DETAILED DESCRIPTION:
This is a Phase 2, single-arm, open, non-randomized, multicenter study of the SINE™ compound selinexor plus low-dose dexamethasone, in combination with bortezomib and daratumumab.

Sixty-two patients with R/R MM who meet eligibility criteria and have none of the exclusion criteria will be enrolled to receive SVDd until either disease progression or intolerance has occurred.

Enrolled patients will take a fixed milligram dose of 100 mg selinexor (on days 1, 8, 15 and 22), plus 40 mg dexamethasone (20 mg IV the day of daratumumab and selinexor and 20 mg oral administration the day after daratumumab and selinexor) both weekly as continuous therapy.

Bortezomib will be given via subcutaneous at dose of 1.3 mg/m2 once weekly on days 1, 8, 15 and 22 during the cycles 1 to cycle 8, and on day 1 and day 15 of each cycle thereafter as continuous therapy.

Daratumumab will be given via intravenous at dose of 16 mg/Kg on days 1, 8, 15 and 22 (weekly) during the cycles 1 and 2, every two weeks (on days 1 and 15) during the cycles 3 to 6 and on day 1 of each cycle thereafter as continuous therapy.

Patients may continue indefinitely and there is no maximum treatment duration

ELIGIBILITY:
Inclusion Criteria:

* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Patient must be at least 18 years of age.
* Patient must have a confirmed diagnosis of symptomatic multiple myeloma and measurable secretory disease, defined as either serum monoclonal protein ≥ 0,5 g/dL or urine monoclonal (light chain) protein ≥ 200 mg/24 hours. For patients in whom measurable disease is performed by serum FLC, the involved FLC should be ≥ 10 mg/dL, with an abnormal serum FLC ratio.
* Patients must have an ECOG performance status of 0, 1 or 2.
* All patients must have received prior treatment with proteasome inhibitors and immunomodulators: A minimum of 2 consecutive cycles of proteasome inhibitors and immunomodulators are required.
* Patients must have received ≥ 3 prior lines of therapy and be refractory to the last line of therapy, or be double refractory to proteasome inhibitors and immunomodulatory drugs on their most recent therapy, regardless of the prior number lines of therapy; or patients were thought to be refractory if they had progressed on or within 60 days of treatment with bortezomib and/or lenalidomide.
* Patient has the following laboratory values within 14 days before Baseline visit (Day 1 of Cycle 1, before study drug administration): Platelet count ≥ 75 x109/L, hemoglobin ≥ 8.0g/dl and absolute neutrophil count (ANC) ≥ 1.5 x 109/L; lower values may be accepted if clearly are due to bone marrow involvement by multiple myeloma (ANC ≥ 1.0 x 109/L and platelets ≥ 50 x109/L if bone marrow infiltration > 60%). Patients receiving hematopoietic growth factor support, including erythropoietin (EPO), darbepoetin, granulocyte-colony stimulating factor (G-CSF) may continue to do so.
* Corrected serum calcium < 14mg/dl.
* Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal, alanine transaminase (ALT): ≤ 2.5 x the upper limit of normal, and total bilirrubin: ≤ 2.0 x the upper limit of normal.
* Calculated creatinine clearance ≥ 20 ml per minute, calculated using the formula of Cockroft and Gault:Multiply times 0.85 if the patient is female, or CrCl >20 mL/min as measured by 24-hour urine collection
* Women of childbearing potential must be practicing a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: eg, established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; barrier methods: condom with spermicidal foam/gel/film/cream/suppository; male partner steritilization (the vasectomized partner should be the sole partner for that subject); true abstinence (when this is in line with the preferred and usual lifestyle of the subject) during and after the study (6 months after the last dose of any component of the treatment regimen).
* A woman of childbearing potential must have a negative serum pregnancy test at screening within 10-14 days and 24 hours before commencing treatment. Females of reproductive potential must commit either to abstain continuously from heterosexual sexual intercourse or to use two methods or reliable birth control simultaneously

Exclusion Criteria:

* Subject has received selinexor or daratumumab therapies previously.
* Patients who are refractory to daratumumab or CD38 targeting antibody.
* Subject has a diagnosis of plasma cell leukemia, primary amyloidosis, monoclonal gammopathy of undetermined significance (MGUS) or smoldering multiple myeloma (SMM).
* Subject has previously received autologous stem cell transplantation within 12 weeks before Cycle Day 1, or has received other anti-myeloma treatment within 2 weeks before Cycle 1 Day 1 (with the exception of an emergency use of a short course [maximum 4 days] of corticosteroids [40 mg/day dexamethasone or equivalent]).
* Subject who had previously received allogeneic stem cell transplantation within the last year or even latter if they have evidence of graft versus host disease.
* Subject has peripheral neuropathy or neuropathic pain grade 2 or higher, as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.
* Subject has had any prior or concurrent invasive malignancy (other than myeloma) within 5 years of study start except adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, localized prostate adenocarcinoma diagnosed ≥ 3 years and without evidence of biochemical failure, or other cancer for which the subject has undergone potentially curative therapy and has no evidence of that disease for ≥ 5 years.
* Subject has had radiation therapy within 28 days of Cycle 1 Day 1.
* Subject has meningeal involvement of multiple myeloma.
* Subject has known severe chronic obstructive pulmonary disease (COPD) (defined as a forced expiratory volume [FEV] in 1 second <60% of predicted normal), persistent asthma, or a history of severe asthma within 5 years. Subjects with known or suspected COPD or asthma must have a FEV test during screening.
* Subjects have known moderate or severe persistent asthma within the past 2 years (see Appendix 8: National Heart, Lung, and Blood Institute (NHLBI) table of asthma severity), or currently has uncontrolled asthma of any classification. (Note that subjects who currently have controlled intermittent asthma or controlled mild ersistene asthma are allowed in the study).
* Unstable cardiovascular function:Symptomatic ischemia, or Uncontrolled clinically-significant conduction abnormalities (e.g., patients with ventricular tachycardia on antiarrhythmics are excluded; patients with 1st degree atrioventricular (AV) block or asymptomatic left anterior fascicular block/right bundle branch block (LAFB/RBBB) will not be excluded), or Congestive heart failure (CHF) of New York Heart Association (NYHA) Class ≥ 3, or Myocardial infarction (MI) within 3 months.
* Patients with uncontrolled hypertension.
* Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose.
* Subject is known to be seropositive for history of human immunodeficiency virus (HIV) or hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg] or antibodies to hepatitis B surface and core antigens [anti HBs and anti-HBc, respectively]) or hepatitis C (anti-HCV antibody positive or HCV-RNA quantitation positive).
* Patients with any GI dysfunction who are unable to swallow tablets, or any GI dysfunction that could interfere with absorption of study treatment
* Serious psychiatric or medical conditions that, in the opinion of the investigator, could interfere with treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Number of responses type to treatment | 1 year
  Note overall response rate (ORR), including stringent complete responses, complete responses (CR), very good partial responses (VGPR), and partial responses (PR) according to the International Myeloma Working Group Criteria (IMWG)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 2 years
  Note incidence of clinical and laboratory toxicities.

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - Hospital Germans Trials i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital ICO de Girona, Girona
  - Hospital ICO de L'hospitalet, L'Hospitalet de Llobregat
  - Hospital 12 de Octubre, Madrid
  - Hospital Clinico de Madrid, Madrid
  - Hospital Morales Meseguer, Murcia
  - Hospital Central de Asturias, Oviedo
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocio, Seville
  - Hospital Dr Peset, Valencia

IPD SHARING:
Plan to Share IPD: No